CLINICAL TRIAL: NCT06525428
Title: A Prospective, Two-cohort Phase II Trial of Standard Systemic Therapy in Combination With High/Low-dose Radiotherapy Plus Toripalimab for Metastatic Colorectal Cancer
Brief Title: Standard Systemic Therapy Combined With High/Low-dose Radiotherapy Plus Toripalimab for Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2024-32-3585
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Microsatellite Stable Metastatic Colorectal Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a first-line cohort A and a second-line cohort B (Experimental)
  Interventions: Drug: standard systemic therapy combined with high/low-dose radiotherapy plus toripalimab

INTERVENTIONS:
Drug: standard systemic therapy combined with high/low-dose radiotherapy plus toripalimab — First-line standard systemic therapies in cohort A include: FOLFOX/XELOX+ bevacizumab, FOLFOX/XELOX+cetuximab (KRAS/NRAS/BRAF WT and left-sided tumors only), FOLFIRINOX+ bevacizumab.
  Second-line standard systemic therapies in cohort B include: FOLFOX/XELOX+ bevacizumab, FOLFOX/XELOX+cetuximab (KRAS/NRAS/BRAF WT), FOLFIRI/irinotecan+raltitrexed/irinotecan/+bevacizumab, FOLFIRI/irinotecan+raltitrexed/irinotecan/+cetuximab (KRAS/NRAS/BRAF WT), based on the previous first-line chemotherapy and adverse events.
  Toripalimab will be given at 240 mg q3w. Radiotherapy regimes include 4-8 fractions of 4-12Gy via SABR or hypofractionated radiotherapy (HFRT) and 5 fractions of 0.5-2Gy via LDRT

SUMMARY:
TORCH-M is a prospective, single-arm, two-cohort, investigator-initiated phase II trial to investigate the efficacy and safety of standard systemic therapy in combination with high/low-dose radiotherapy plus toripalimab in paitents with microsatellite stable metastatic colorectal cancer (MSS mCRC). Eligible patients will be assigned to two cohorts according to previous treatment: a first-line cohort A and a second-line cohort B. Patients in both arms will first receive one cycle of standard systemic therapy and toripalimab, followed by high/low-dose radiotherapy, and then continue with standard systemic therapy and toripalimab.The survival benefits, response rates, and adverse effects will be analyzed.

DETAILED DESCRIPTION:
First-line standard systemic therapies in cohort A include: FOLFOX/XELOX+ bevacizumab, FOLFOX/XELOX+cetuximab (KRAS/NRAS/BRAF WT and left-sided tumors only), FOLFIRINOX+ bevacizumab.

Second-line standard systemic therapies in cohort B include: FOLFOX/XELOX+ bevacizumab, FOLFOX/XELOX+cetuximab (KRAS/NRAS/BRAF WT), FOLFIRI/irinotecan+raltitrexed/irinotecan/+bevacizumab, FOLFIRI/irinotecan+raltitrexed/irinotecan/+cetuximab (KRAS/NRAS/BRAF WT), based on the previous first-line chemotherapy and adverse events.

Toripalimab will be delivered at 240 mg q3w. Radiotherapy regimes include 4-8 fractions of 4-12Gy via SABR or hypofractionated radiotherapy (HFRT) and 5 fractions of 0.5-2Gy via LDRT.

ELIGIBILITY:
Inclusion Criteria:

Age between18 and 75 years old.

An Eastern Cooperative Oncology Group (ECOG) performance status ≤1.

Histopathological confirmed MSS/pMMR adenocarcinoma of the colon or rectum.

At least one evaluable metastatic lesion for radiotherapy and evaluation according to RECIST 1.1.

Treatment naive (first-line cohort) and progressed on after first-line therapy or stopped first-line therapy due to unacceptable toxic effects (second-line cohort).

Prior radiotherapy completed at least 4 weeks before enrollment.

Adequate bone-marrow, hepatic, and renal function: neutrophils ≥ 1.5 × 10^9/L, Hb ≥ 90 g/L, PLT ≥ 100 × 10^9/L, ALT/ AST≤2.5 ULN, Cr≤1 ULN.

Sign the informed consent and have good compliance.

Exclusion Criteria:

Neutrophil < 1.5×10^9/L, PLT < 100×10^9/L (PLT < 80×10^9/L in patients with liver metastasis), or Hb < 90g/L; blood transfusion within 2 weeks before enrollment is not allowed to meet the enrollment criteria.

TBIL > 1.5 ULN, or TBIL > 2.5 ULN in patients with liver metastasis. AST or ALT > 2.5 ULN, or ALT and / or AST > 5 ULN in patients with liver metastasis.

Cr > 1.5 ULN, or creatinine clearance < 50ml / min (calculated according to Cockcroft Gault formula).

APTT > 1.5 ULN, PT > 1.5 ULN (subject to the normal value of the clinical trial research center).

Serious electrolyte abnormalities. Urinary protein ≥ 2+, or 24-hour urine protein ≥1.0g/24h. Uncontrolled hypertension: SBP >140mmHg or DBP > 90mmHg. The presence of gastrointestinal diseases such as gastric or duodenal active ulcers, ulcerative colitis or unresected tumours with active bleeding; or other conditions likely to cause gastrointestinal bleeding or perforation; or unhealed gastrointestinal perforation or gastrointestinal fistula after surgical treatment.

A history of arterial thrombosis or deep vein thrombosis within 6 months; a history of bleeding or evidence of bleeding tendency within 2 months.

A history of heart disease within 6 months (including congestive heart failure, acute myocardial infarction, severe/unstable angina, coronary artery bypass grafting, cardiac insufficiency ≥ NYHA grade 2 and LVEF<50%).

Uncontrolled malignant pleural effusion, ascites, or pericardial effusion. History of anti-PD-1, PD-L1, PD-L2, CTLA-4 or any other specific T cell co-stimulation or checkpoint pathway targeted therapy.

The presence of a clinically detectable second primary malignancy, or history of other malignancies within 5 years excluding adequately treated non-melanoma skin cancer, carcinoma in situ of cervix and superficial bladder tumour (non-invasive tumour, or carcinoma in situ, or T1).

A history of liver disease including, but not limited to HBV infection or HBV DNA positive(≥1×10^4/ml), HCV infection or HCV DNA positive(≥1×10^3/ml) and liver cirrhosis.

Pregnant or lactating women or women who may be pregnant have a positive pregnancy test before the first medication; Or the female participants themselves and their partners who were unwilling to implement strict contraception during the study period.

The investigator considers that the subject is not suitable to participate in this clinical study due to any clinical or laboratory abnormalities or compliance problems.

Serious mental abnormalities. The diameter of brain metastasis is greater than 3cm or the total volume is greater than 30cc.

Clinical or radiological evidence of spinal cord compression, or tumours within 3 mm of the spinal cord on MRI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 2 years
  Defined as the time from initiation of treatment to PD or death from any cause.

SECONDARY OUTCOMES:
OS | Up to 3 years
  Defined as the time from initiation of treatment to death from any cause.
ORR | Up to 1 year
  The percentage of patients with objective response in all metastatic lesions.
DCR | Up to 1 year
  The percentage of patients with disease control in all metastatic lesions. Disease control is defined as CR, PR, or stable disease (SD) per RECIST v1.1 and iRECIST after treatment.
Adverse events | Up to 3 years
  The percentage of patients with treatment-related acute toxicities as assessed by NCI CTCAE v5.0, from treatment initiation until 90 days upon completion of immunotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China